CLINICAL TRIAL: NCT05440695
Title: Can We Detect Hypotension Episodes That Were Not Identified in the Non-Invasive Blood Pressure During Cesarean Section? A Randomized Controlled Trial
Brief Title: Undetectable Hypotension Episodes in Cesarean Section
Status: Completed | Type: Observational
Sponsor: Asude AYHANt (Other)
Responsible Party: Sponsor-Investigator, Asude AYHANt, Assistant Professor of Anaethesiology and Reanimation, Baskent University
Organization: Baskent University (Other)
Other Study IDs: KA13/33
Record Dates: First submitted 2022-06-08; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Pregnancy Related; Anesthesia; Blood Pressure
Keywords: Anesthesia; Obstetrical; Cesarean section; Arterial pressure; Blood pressure; Newborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- CNAP Group: The CNAP finger cuff and NIBP cuff were on the same arm of the patient while the intravenous catheter was on the contralateral side. After intrathecal injection, systolic, diastolic, and mean blood pressures were measured and were recorded manually at every minute on the CNAP monitor.
  Interventions: Device: Continuous non-invasive arterial pressure (Infinity® CNAPTM, Dräger)
- NIBP Group: In the control group, only oscillometric NIBP measurements were done in pregnant women similar to the study group without a CNAP. After intrathecal injection, systolic, diastolic, and mean blood pressures with oscillometric method were set at the frequency of 3 minutes for the first 15 minutes, and at 5-minute intervals thereafter, and were recorded manually.

INTERVENTIONS:
Device: Continuous non-invasive arterial pressure (Infinity® CNAPTM, Dräger) — The basic working principle of CNAP is to keep the blood volume of the finger arteries constant by applying an exterior pressure to the vessel wall, that is done by an electronic system controlling the pressure inside a cuff around the finger. The pressure in the cuff, which is needed to keep the volume constant during arterial pulsation, corresponds to the AP.
  Groups: CNAP Group

SUMMARY:
In order to evaluate the efficacy and necessity of continuous non-invasive arterial pressure (CNAP) by comparing it with non-invasive blood pressure (NIBP) in order to understand whether it has advantages over oscillometric technique for detection of hypotensive episodes in healthy pregnant women who underwent cesarean section (C/S) under neuraxial anesthesia. This prospective study will evaluate healthy pregnant women at term, who were scheduled for elective C/S under spinal anesthesia. Subjects were randomly assigned into 2 groups to receive either CNAP and NIBP or only NIBP. A thirty percent decrease in systolic blood pressure from either baseline or the measured values in the first two minutes, or if the systolic blood pressure was less than 90mmHg, is considered hypotension. Pre-, peri- and post-operative specifications, newborn characteristics, and complications were recorded and compared.

DETAILED DESCRIPTION:
The aim of the study was to test the hypothesis that whether continuous non-invasive arterial pressure (CNAP) is able to identify the hypotensive episodes that were not disclosed (or identified) in the non-invasive blood pressure (NIBP), or, detects earlier compared to NIBP in healthy pregnant women who underwent C/S under neuraxial anesthesia. We also evaluated the association between monitoring CNAP vs NIBP and outcomes as a secondary endpoint.

At least 40 participants were planned to be included in each arm, considering the unforeseen technical problems (in accordance with the "Power and Sample Size Program", the inclusion of at least 29 patients was necessary for both groups for a power 0.80, alpha 0.05 and a standard deviation of 0.04).

Healthy pregnant women at term, who were scheduled for the elective C/S under spinal anesthesia in an academic tertiary care unit between February 2014 and February 2015, comprised the study group. The exclusion criteria for the study were; 1) emergency C/S, 2) simultaneous gynecological interventions with C/S such as myomectomy, tubal ligation, placental abnormalities, etc., 3) if C/S was performed in failure of labor to progress, 4) the presence of any systemic disease, 5) preeclampsia or eclampsia, 6) drug hypersensitivity - for the ones that are used in the C/S -, 7) multiple pregnancies, 8) those pregnancies with any intrauterine fetal pathology, and 9) more than two missing consecutive NIBP readings.

Subjects were randomly assigned into 2 groups to receive either CNAP and NIBP or only NIBP. CNAP finger cuff (Infinity® CNAPTM, Dräger) was used for calibrate the device before the first measurement then calibration was repeated every 30 minutes.

In the CNAP group, the CNAP finger cuff and NIBP cuff were on the same arm of the patient while the intravenous catheter was on the contralateral side. In the control group, only oscillometric NIBP measurements were done in pregnant women similar to the study group without a CNAP.

After intrathecal injection, systolic, diastolic, and mean blood pressures were measured and were recorded manually at every minute on the CNAP monitor, and the oscillometric NIBP measurements were set at the frequency of 3 minutes for the first 15 minutes, and at 5-minute intervals thereafter, and were recorded manually.

Demographic and pregnancy-related characteristics (age, parity, gravidas of the pregnant women, weeks of gestation, and the type of fertilization [spontaneous or in vitro fertilization (IVF)] were recorded.

All parturients underwent C/S after 8 hours of fasting period without any pharmacological premedication. They were monitored with 5 lead electrocardiograms, and pulse oximetry in the operating theater. By providing the monitorization, a total of 1000ml of Ringer's lactate infusion was given by an intravenous line with an 18-gauge cannula as pre-load/co-load. A 12.5 mg of hyperbaric bupivacaine was administered to all pregnant women in the left lateral decubitus position with a 26-gauge atraumatic spinal needle at the L3-4 or L4-5 interval. After the spinal injection, the patients were placed in a supine position, and the uterus was directed to the left side by using a support under the right hip. Oxygen was given to all the parturients at 3 lt / min by nasal cannula.

The block-level was assessed by loss of sensitivity to cold. When it reached the T4 skin dermatome, the surgery was started. Motor block was determined and recorded using the modified Bromage scale (0 = no block, 1 = knee flexion possible, leg unable to lift, 2 = ankle flexion and finger movements possible, unable to move the knee, 3 = full motor block in the lower extremity). The sensitivity to cold was checked every 5 minutes and the maximum block level was recorded. Analgesia was evaluated using a visual analog scale scorer (0 = no pain, 10 = most severe pain). Time from intrathecal injection to delivery (block-delivery time), time from skin incision to delivery (skin-birth time), time from uterine incision to delivery (uterus-delivery time) were recorded.

After the baby was born, the mother was sedated with midazolam 0.03 mg/kg so that the Ramsay sedation score was 2, and analgesia was provided with fentanyl 0.5 μg/kg if necessary. As the umbilical cord was clamped, 2g of cephalosporin and 5 IU of oxytocin were administered intravenously, and 15 IU oxytocin in 1000 ml Ringer's lactate was infused in an hour.

Peri/Post-Operative Periods Patients with a thirty percent decrease in systolic blood pressure from either baseline or the measured values in the first two minutes, or with systolic blood pressure less than 90mmHg; which is considered as hypotension (13), were treated with a bolus of 200 ml Ringer's lactate solution. If blood pressure did not improve after 3 minutes, 5 mg intravenous ephedrine was administered.

A decrease in heart rate below 50 beats/min was considered as bradycardia, and 0.5mg intravenous atropine was administered when encountered.

The nausea-vomiting score was calculated as follows; the absence of nausea -0, nausea without vomiting -1, and vomiting -2 points.

Patient discomfort for non-invasive blood pressure cuff and CNAP cuff scored was as 0, 1, 2, and 3 for; no discomfort, mild discomfort, moderate discomfort, and severe discomfort, respectively.

The amount of administered intravenous fluids and ephedrine during anesthesia, the umbilical artery blood gas values, and APGAR scores at 1st minute, and at 5th minutes were also recorded.

Complications, ie, postoperative fever, bleeding, need a transfusion for blood and blood products, aspiration, atelectasis, and postspinal headache, were noted at the postoperative 24th and 48th hours. The length of stay hospital stay for the mother and baby, the requirement for intensive care unit, and/or mechanical ventilator were assessed, separately.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at term, who were scheduled for the elective (planned) C/S under spinal anesthesia

Exclusion Criteria:

* emergency C/S,
* simultaneous gynecological interventions with C/S such as myomectomy, tubal ligation, placental abnormalities, etc.,
* C/S that was performed in failure of labor to progress,
* the presence of any systemic disease,
* preeclampsia or eclampsia,
* hypersensitivity to drugs that are used in C/S,
* multiple pregnancies,
* pregnancies with any intrauterine fetal pathology,
* cases with more than two missing consecutive NIBP readings.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study group consisted of pregnant women at term, who were scheduled for the elective (planned) C/S under spinal anesthesia in an academic tertiary care unit. Subjects were randomly assigned into 2 groups to receive either CNAP and NIBP or only NIBP.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
Detection of hypoptensive episodes | Approximately 100minutes/patient (till the end of the C/S).
  Hypotensive

SECONDARY OUTCOMES:
The association between monitoring CNAP vs NIBP and other related outcomes - Anesthesia time to reach T4 level | Approximately 100minutes/patient (till the end of the C/S).
  Anesthesia time to reach T4 level (minutes)
The association between monitoring CNAP vs NIBP and other related outcomes - Skin incision time (minutes) | Approximately 100minutes/patient (till the end of the C/S).
  Skin incision time (minutes)
The association between monitoring CNAP vs NIBP and other related outcomes - Uterine incision time (minutes) | Approximately 100minutes/patient (till the end of the C/S).
  Uterine incision time (minutes)
The association between monitoring CNAP vs NIBP and other related outcomes - Time to leave the operating theater (minutes) | Approximately 100minutes/patient (till the end of the C/S).
  Time to leave the operating theater (minutes)
The association between monitoring CNAP vs NIBP and other related outcomes - Intraoperative fluid (ml) | Approximately 100minutes/patient (till the end of the C/S).
  Intraoperative fluid (ml)
The association between monitoring CNAP vs NIBP and other related outcomes - The need and amount of ephedrine used | Approximately 100minutes/patient (till the end of the C/S).
  The need (number of patients) and amount (mg) of ephedrine used
The association between monitoring CNAP vs NIBP and other related outcomes - Bolus of 200 ml Ringer's lactate solution | Approximately 100minutes/patient (till the end of the C/S).
  The need (number of patients) of bolus 200 ml Ringer's lactate solution
The association between monitoring CNAP vs NIBP and other related outcomes - Nausea | After C/S - early postoperative period - through study completion, an average of 1 year
  Nausea (number of patients)
The association between monitoring CNAP vs NIBP and other related outcomes - Vomiting | After C/S - early postoperative period - through study completion, an average of 1 year
  Vomiting (number of patients)
The association between monitoring CNAP vs NIBP and other related outcomes - Length of Hospitalization (days) | Length of Hospitalization - through study completion, an average of 1 year
  Length of Hospitalization (days)
The association between monitoring CNAP vs NIBP and other related outcomes - Cuff discomfort | Approximately 100minutes/patient (till the end of the C/S).
  Cuff discomfort (Scale based: No - Mild - Moderate or Severe)
The association between monitoring CNAP vs NIBP and other related outcomes - Newborns' Blood Gas Analysis | At the time of birth - through study completion, an average of 1 year
  Newborns' Blood Gas Analysis - Umblical Artery pH
The association between monitoring CNAP vs NIBP and other related outcomes - Newborns' Blood Gas Analysis | At the time of birth - through study completion, an average of 1 year
  Newborns' Blood Gas Analysis - Umblical Artery pO2
The association between monitoring CNAP vs NIBP and other related outcomes - Newborns' Blood Gas Analysis | At the time of birth - through study completion, an average of 1 year
  Newborns' Blood Gas Analysis - Umblical Artery pCO2
The association between monitoring CNAP vs NIBP and other related outcomes - Newborns' Blood Gas Analysis | At the time of birth - through study completion, an average of 1 year
  Newborns' Blood Gas Analysis - Umblical Artery Lactate
The association between monitoring CNAP vs NIBP and other related outcomes - Newborns' APGAR score | After birth at 1st minute
  Newborns' APGAR score
The association between monitoring CNAP vs NIBP and other related outcomes - Newborns' APGAR score | After birth at 5th minutes
  Newborns' APGAR score

CONTACTS AND LOCATIONS:
Overall Officials: Aynur C FIRAT, M.D., Principal Investigator — Baskent University School of Medicine, Department of Anaesthesiology and Reanimation

IPD SHARING:
Plan to Share IPD: Yes
When the study is completed and totally shaped out as an academic manuscript, the individual participant data (IPD) will be available to other researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available when the related manuscript is published in a scientific journal. So, the researchers will be able to reach the manuscript whenever they want-upon the regulations of the published journal.
Access Criteria: Access will be done throughout the journal's website or digital object identifier system (DOI).

REFERENCES:
- [Background] Ngan Kee WD. Prevention of maternal hypotension after regional anaesthesia for caesarean section. Curr Opin Anaesthesiol. 2010 Jun;23(3):304-9. doi: 10.1097/ACO.0b013e328337ffc6. PMID 20173633
- [Result] Ilies C, Bauer M, Berg P, Rosenberg J, Hedderich J, Bein B, Hinz J, Hanss R. Investigation of the agreement of a continuous non-invasive arterial pressure device in comparison with invasive radial artery measurement. Br J Anaesth. 2012 Feb;108(2):202-10. doi: 10.1093/bja/aer394. Epub 2011 Dec 12. PMID 22171358
- [Result] Ilies C, Kiskalt H, Siedenhans D, Meybohm P, Steinfath M, Bein B, Hanss R. Detection of hypotension during Caesarean section with continuous non-invasive arterial pressure device or intermittent oscillometric arterial pressure measurement. Br J Anaesth. 2012 Sep;109(3):413-9. doi: 10.1093/bja/aes224. Epub 2012 Jul 12. PMID 22798273
- [Result] Gupta D, Soskin V, Marjanovic M, Amhaz H, Mazumdar A. CONTINUOUS NON-INVASIVE ARTERIAL PRESSURE DEVICE AS AN ADJUNCT TO RECOGNIZE FLUCTUATING BLOOD PRESSURES DURING ELECTIVE CESAREAN SECTION UNDER SUBARACHNOID BLOCKADE (SAB). Middle East J Anaesthesiol. 2016 Feb;23(4):385-400. PMID 27382807
- [Result] Hahn R, Rinosl H, Neuner M, Kettner SC. Clinical validation of a continuous non-invasive haemodynamic monitor (CNAP&trade; 500) during general anaesthesia. Br J Anaesth. 2012 Apr;108(4):581-5. doi: 10.1093/bja/aer499. Epub 2012 Feb 3. PMID 22307242